CLINICAL TRIAL: NCT04242836
Title: Development and Validation of a Computer-based Digital Near-vision Optotype Based on the Greek Version of the Print MNREAD.
Brief Title: Development and Validation of a Digital Optotype for Near Vision in Greek Language.
Acronym: DeDART
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Associate Professor of Ophthalmology, Democritus University of Thrace
Other Study IDs: ES3/Th2/27-03-2019
Record Dates: First submitted 2020-01-08; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Presbyopia; Low Vision; Near Vision
Keywords: digital near vision chart; critical print size; reading acuity; reading speed; digital Greek MNREAD
MeSH Terms: conditions — Presbyopia; Vision, Low; Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: 1. 70 patients with normal vision (NVG) with adequate literacy of written Greek language
  2. 30 patients with low vision (LVG) with adequate literacy of written Greek language
  These patients are tested on the printed Greek MNREAD
  Interventions: Diagnostic Test: MNREAD testing
- Study group: The same patients as those in the control group (NVG, LVG) are tested on the digital version of the Greek MNREAD (DeDART)
  Interventions: Diagnostic Test: MNREAD testing

INTERVENTIONS:
Diagnostic Test: MNREAD testing — One randomly selected eye is included for each study participant. Participants respond to the near vision chart with defined environmental circumstances at 40cm viewing distance. All four parameters (RA, MRS, CPS and ACC) are evaluated.

SUMMARY:
Primary objective of our study is to develop and validate a computer-based digital near-vision optotype based on the Greek version of the print MNREAD.

DETAILED DESCRIPTION:
Present study aims to develop and validate a computer-based digital near-vision optotype based on the Greek version of the print MNREAD.

Specifically, it aims to evaluate the level of agreement between the conventional printed greek MNREAD chart and the corresponding digital chart, as well as test-retest reliability of the digital optotype.

To address these aims, four reading parameters measured with the print and the digital version are compared. These parameters are the following:

1. Reading Acuity (RA)
2. Maximum Reading Speed (MRS)
3. Critical Print Size (CPS)
4. Accessibility Index (ACC)

All the comparisons take place in two groups: a) a Normal Vision Group (NVG), and b) a Low Vision Group (LVG) in order to estimate the reading capacity in a population with a wide range of vision.

ELIGIBILITY:
Inclusion Criteria:

* adequate literacy of written Greek language

Exclusion Criteria:

* dyslexia
* attention-deficiency
* former diagnosis of mental diseases
* former diagnosis of psychiatric diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal- and low-sighted participants aged 18 to 75 years
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Reading Acuity (RA) | through study completion, an average of 8 months
  The smallest print that the patient can read without making significant errors, and can be calculated by the following formula:
  Acuity (in logMAR)= 1.4 - (sentences x 0.1) + (errors x 0.01).
Maximum Reading Speed (MRS) | through study completion, an average of 8 months
  The patient's reading speed when reading is not limited by print size , and is calculated by averaging the speed of the sentences with print size larger than the CPS. [(in words per minute (wpm)]
Critical Print Size (CPS) | through study completion, an average of 8 months
  The smallest print size at which patients can read with their MRS, and is identified as the print size of the sentence fulfilling this criterion: all of the following sentences are read at a speed that is 1.96 times the standard deviation below the average of the larger preceding sentences (that is the MRS). In other words, it is defined as the smallest print size that yields 90% of the MRS [(in logMAR)]
Accessibility Index (ACC) | through study completion, an average of 8 months
  The mean reading speed measured across the 10 largest print sizes (1.3 to 0.4 logMAR) of the MNREAD Acuity Chart at 40 cm normalized by 200 wpm, which was the mean value for a group of 365 normally sighted young adults aged 18 to 39 years old.

SECONDARY OUTCOMES:
Intraclass Correlation Coefficients (ICCs) for study participants | through study completion, an average of 8 months
  Level of agreement between the print and the digital version are evaluated by calculation of the ICCs for the 4 reading parameters (RA, MRS, CPS, ACC).
Test-retest Intraclass Correlation Coefficients (ICCs) | through study completion, an average of 8 months
  Test-retest reliability of the digital optotype is evaluated by ICCs for the 4 reading parameters (RA, MRS, CPS, ACC)..

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (1):
- University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

REFERENCES:
- [Derived] Labiris G, Panagiotopoulou EK, Chatzimichael E, Tzinava M, Mataftsi A, Delibasis K. Introduction of a digital near-vision reading test for normal and low vision adults: development and validation. Eye Vis (Lond). 2020 Oct 22;7:51. doi: 10.1186/s40662-020-00216-0. eCollection 2020. PMID 33102611